CLINICAL TRIAL: NCT01810367
Title: ABX Combined With Cisplatin Compared With Gemcitabine Combined With Cisplatin in First Line Treatment of Locally Advanced or Metastatic Non-small Cell Lung Cancer Stage II Randomized Controlled Trials
Brief Title: ABX Combined With Cisplatin Compared With Gemcitabine Combined With Cisplatin in NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Chang Jian Hua, Vice director of department of chemotherapy, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABX-CJH
Record Dates: First submitted 2013-03-11; First posted 2013-03-13 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Non Small Cell Lung Cancer
Keywords: PFS
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ABX Combined With Cisplatin (Experimental): ABX，100mg/m2，d1、8、15，ivgtt,in 30 min，28day one cycle； cisplin 75mg/m2 d1 ivgtt
  Interventions: Drug: ABX Combined With Cisplatin
- Gemcitabine Combined With Cisplatin (Active Comparator): gemcitabine 1000mg/m2，d1、8；cisplatin 75mg/m2 d1 ivgtt,3 weeks one cycle.
  Interventions: Drug: Gemcitabine Combined With Cisplatin

INTERVENTIONS:
Drug: ABX Combined With Cisplatin
  Arms: ABX Combined With Cisplatin
Drug: Gemcitabine Combined With Cisplatin
  Arms: Gemcitabine Combined With Cisplatin

SUMMARY:
Assess the PFS/ORR/OS of ABX Combined With Cisplatin Compared With Gemcitabine Combined With Cisplatin in first Treatment of NSCLC

ELIGIBILITY:
1.18~75 years 2.Patients who were diagnosed by the histologic, cytologic diagnosis of IIIb-IV non-small cell lung cancer 3.Presence of at least one index lesion measurable by CT scan or MRI 4.Ecog0-1 5.Expected life time longer than 12 weeks 6.Normal laboratory values:

* leucocyte ≥ 4×109/L
* neutrophil ≥ 1.5×109/L
* platelet ≥ 100×109/L
* Hemoglobin ≥ 10g/L
* ALT and
* AST ≤ 2.5×ULN (≤ 5×ULN if liver metastasis) 7.Signed written informed consent

Exclusion Criteria:

* Patients have used drugs according to protocol
* Patients were allergic to pemetrexed or cisplatin
* Patients received radiotherapy or other biological treatment 4 weeks before the trial
* Uncontrolled hydrothorax or hydropericardium
* neuropathy toxicity ≥ CTC 3
* Severe symptomatic heart disease
* Active upper gastrointestinal ulcer or digestive disfunction
* Severe infection or metabolic disfunction
* Patients with other malignant tumor
* Uncontrolled brain metastases
* Patients have accepted other clinical trials
* Female patients during their pregnant and lactation period, or patients without contraception

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2011-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
PFS | from the first cycle of treatment (day one) to two month after the last cycle

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer hospital Fudan University, Shanghai, Shanghai Municipality, China